CLINICAL TRIAL: NCT04326452
Title: The Use of a Bidirectional Oxygenation Valve in the Management of Respiratory Failure Due to COVID-19 Infection
Brief Title: Treating COVID-19 With a Bidirectional Oxygenation Valve
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: TMC HealthCare (Other)
Collaborators: PEEP Medical, LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: COVID19PEEP2020; GO2 PEEP Study (Other: GO2 Devices)
Record Dates: First submitted 2020-03-25; First posted 2020-03-30 (Actual); Last update posted 2022-05-04 (Actual); Status verified 2020-03

CONDITIONS: Coronavirus Infection
MeSH Terms: conditions — Coronavirus Infections

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Enrolled Subjects (Experimental): The purpose of this study is to compare the use of our bidirectional oxygenation mouthpiece with conventional oxygen support versus conventional oxygen support of any Person Under Investigation for infection by the COVID-19 virus.
  Interventions: Device: bidirectional oxygenation mouthpiece

INTERVENTIONS:
Device: bidirectional oxygenation mouthpiece — Use of our bidirectional oxygenation mouthpiece with conventional oxygen support.

SUMMARY:
This study will utilize a single center internal control study design. The objective of this study is to determine the feasibility and safety of a bidirectional oxygenation PEEP generating mouthpiece when combined with oxygen by non-rebreather face mask, compared to support by oxygen non-rebreather face mask alone.

DETAILED DESCRIPTION:
We have developed a simple and straightforward silicone rubber-made oral appliance that promotes positive expiratory airway pressures with the potential to enhance respiratory function while preventing and reversing atelectasis and hypoxia. The purpose of this study is to compare the use of our bidirectional oxygenation mouthpiece with conventional oxygen support versus conventional oxygen support of any Person Under Investigation for infection by the COVID-19 virus.

ELIGIBILITY:
Inclusion Criteria:

* Oxygen saturation <93%
* Able to provide informed consent
* Not currently requiring intubation
* Receiving oxygen by face mask

Exclusion Criteria:

* Unable or unwilling to provide informed consent, cognitive impairment
* Rapidly decompensating status requiring urgent or emergent higher level of care

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2020-03-27 (Actual); Primary Completion 2021-03-27 (Actual); Study Completion 2021-03-27 (Actual)

PRIMARY OUTCOMES:
Pulse oximetry level | Change from Baseline pulse oximetry level at 15 minutes post treatment
  The primary endpoint for this feasibility study is pulse oximetry level after treatment with a Bidirectional Oxygenation Valve

SECONDARY OUTCOMES:
Respiratory rate | Change from Baseline clinical measurements at 15 minutes post treatment
Heart rate | Change from Baseline clinical measurements at 15 minutes post treatment
Blood pressure | Change from Baseline clinical measurements at 15 minutes post treatment
Systemic carbon dioxide | Change from Baseline clinical measurements at 15 minutes post treatment
  Venous and arterial blood gases, if available, will be combined to report systemic carbon dioxide.

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - TMC HealthCare, Tucson, Arizona
  - Stanford University, Stanford, California
  - Emory Saint Joseph's Hospital, Atlanta, Georgia